CLINICAL TRIAL: NCT04354324
Title: Treatment Efficacy and Safety of Low-dose Radioiodine Ablation for Intermediate-risk Differentiated Thyroid Carcinoma Patients Without Metastasis: a Double-blind Randomized Clinical Trial
Brief Title: Treatment Efficacy and Safety of Low-dose Radioiodine Ablation for Intermediate-risk Differentiated Thyroid Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Huijuan Feng, Deputy chief physician, Zhujiang Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-KY-050-02
Record Dates: First submitted 2020-03-01; First posted 2020-04-21 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Papillary Thyroid Cancer
Keywords: Radioactive iodine; Papillary thyroid carcinoma
MeSH Terms: conditions — Thyroid Cancer, Papillary | interventions — Iodine-131

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The test group (Experimental): Oral administration of 30mci once on an empty stomach.
  Interventions: Drug: Radioiodine
- The control group (Active Comparator): Oral administration of 100mci once on an empty stomach.
  Interventions: Drug: Radioiodine

INTERVENTIONS:
Drug: Radioiodine — The test group: low dosage (30mci). The control group: high dosage (100mci).
  Other Names: 131 I

SUMMARY:
Primary objective: The 3-years disease-free survival was compared between low-dose group (30 mCi) and high-dose group (100 mCi).

Secondary objective: The successful remnant ablation, efficacy, 3-year progression-free survival and safety were compared between low-dose group (30 mCi) and high-dose group (100 mCi).

Research Hypothesis：The 3-year disease-free survival of low-dose group (30mci) may not be lower than that of high-dose group (100 mci) in intermediate-risk thyroid papillary carcinoma patients with no structural or functional lesions and stimulated thyroglobulin(ps-Tg)1-20ng/ml.

Study design：Single-center, randomized, double-blinded Sample size：254 patients Follow-up：The measurement of serum thyroid function, thyroglobulin/ anti-thyroglobulin antibody(Tg/TgAb) and neck ultrasonography were performed every 3-12 months during the 3 years according to patients' condition, and computerized tomography(CT) scan, positron emission tomography/computed tomography(PET/CT) and diagnostic whole-body 131I scan were added if necessary. Intervention：Randomly allocated into two groups to receive either 30 mCi (low-dose group) or 100 mCi (high-dose group ) radioiodine for post-thyroidectomy ablation therapy.

Evaluation index：Primary evaluation index: The 3-year disease-free survival. Secondary evaluation index: Successful remnant ablation, efficacy, the 3-year progression-free survival and safety.

DETAILED DESCRIPTION:
Intermediate risk papillary thyroid carcinoma(PTC) patients with no structural and functional lesions and stimulated thyroglobulin( s-Tg) 1-20ng/ml were randomly divided into low-dose group (30 mCi) and high-dose group (100 mCi). The 3-years disease-free survival was compared between two groups.The successful remnant ablation, efficacy, 3-year progression-free survival and safety (short-term and long-term adverse reactions) were compared between two groups (30mci, 100mci).The 3-year disease-free survival of low-dose group (30mci) may not be lower than that of high-dose group (100mci) in intermediate-risk thyroid papillary carcinoma patients with no structural or functional lesions and stimulated thyroglobulin 1-20ng/ml.This study is a single-center, randomized, double-blind parallel controlled study initiated by Southern Medical University. The follow-up period was 3 years.The study was divided into two groups: the test group (30mci) and the control group (100mci). And the subjects were randomly assigned to the test group or the control group. This study is a double-blind trial. The specification of the outer packaging of the control drug is the same as that of the test drug, and the subjects are blinded. According to literature reports and pre-clinical data, the disease-free survival of the control group was 92%, non-inferiority cutoff value was δ = 7%, A total of 254 subjects are generated from a=0. 025 (one-sided test), Power=0.8, proportion=0.5(control group) and lost rate =10% (two groups) by Power Analysis and Sample Size(PASS) software. Patients admitted to the department for 131I therapy are recruited by means of propaganda, science popularization and so on. A total of 254 patients with PTC were enrolled in the study which was conducted in the Nuclear Medicine Department, Zhujiang Hospital of Southern Medical University from June 2019 to June 2024. The test group: low dosage (30mci).The control group: high dosage (100mci).The name, appearance and packaging of the test group and the control group are the same, the dosage forms are different, but participants can be made into the same volume. Therefore, the products of two groups can not be distinguished with the naked eye but measuring instruments. Subjects must be screened within one week before random enrollment. The informed consent of the patient will be obtained after a detailed explanation of the study to each subject and before any screening process or evaluation.

During the screening visit, the following procedures will be carried out / the following information will be collected:

Demographic characteristics (Include date of birth, gender and race); Medical and treatment history; Operation and postoperative pathology; Vital signs（breath/ pulse /blood pressure/ pulse rate）; Physical examination; Lab examination (hematology/biochemistry/urinalysis); Thyroid function test; Tg / TgAb; Tumor markers; Pregnancy test (fertile women); 12-Lead Electrocardiogram; Neck ultrasonography; CT of neck and chest; 131I whole-body scan; Neck MRI (not-required item, performed when neck ultrasonography suggests suspicious lymph nodes but can not be diagnosed).

Combined medications and adverse events record Treatment Stage 1(V2,0) Vital signs（breath/ pulse /blood pressure/ pulse rate）; Physical examination; Lab examination (hematology/biochemistry/urinalysis); Thyroid function test; Tg/TgAb; 12-Lead Electrocardiogram; Neck ultrasonography; 131I whole-body scan; Combined medications and adverse events record. Following Stage(V(n+1),8 weeks±n day（s)） Lab examination (hematology/biochemistry/urinalysis); Thyroid function test; Tg/TgAb; Tumor markers; Neck ultrasonography; CT of neck and chest; 131I whole-body scan; Neck MRI (not a necessary item, performed when neck ultrasonography suggest suspicious lymph nodes but can not be diagnosed); PET/CT(not a necessary item,performed when stimulated thyroglobulin >10ng/ml and 131I whole body scan negative) Combined medications and adverse events record. Observation Index

(1) Effectiveness observation Index: disease-free survival, successful remnant ablation, efficacy, Progression-free survival

1. Primary observation Index: That is the Percentage of patients who achieve excellent response in the 3-year follow-up period in the study.
2. Secondary observation Index: Successful remnant ablation, efficacy, Progression-free survival.

Successful remnant ablation: Subjects evaluated at 6-12 months after the initiation of treatment met one of the following two conditions: 1) absence radioactive iodine uptake in the thyroid bed according to a diagnostic 131I whole-body scan. 2) Serum stimulated thyroglobulin was <1 ng/ml or suppressed thyroglobulin was <0.2 ng/ml.

Efficacy: Excellent response, Intermediate response, Biochemical incomplete response, Structural incomplete response.

Progression-free survival: Subjects met any one of the following conditions: 1) functional or structural lesions appeared during follow-up; 2) When sTg> 1 ng/ml or suppressed Tg> 0.2 ng/ml, the serum Tg level increased by more than 25% compared to the previous;3)TgAb was negative at the time of enrollment, and it was positive and persistently elevated during follow-up. The others were defined as progression-free survival.

(2)Safety index: Incidence of short-term and long-term adverse reactions after 131I treatment(time points to distinguish short-term and long-term is 3months ) are listing in table 2, which includes gastrointestinal side effect, radiation thyroiditis, salivary adenitis, myelosuppression, secondary cancer, etc.

Observation time point Patients return to our hospital every 3-12 months to be performed neck ultrasound and thyroid function, Tg / TgAb and other tests, if it is necessary, neck and chest CT, diagnostic 131I whole body imaging, or PET / CT were performed according to patients'condition.

Evaluation Index Primary Evaluation Index Disease-free survival, defined as the Percentage of patients who achieve excellent response in the 3-year follow-up period in the study.

Secondary Evaluation Index

1. Effectiveness Evaluation Index: successful remnant ablation, efficacy,progression-free survival
2. Safety Index: Incidence of short-term and long-term adverse reactions after 131I treatment(time points to distinguish short-term and long-term is 3months )，which includes gastrointestinal side effect, radiation thyroiditis, salivary adenitis, myelosuppression, secondary cancer, etc.
3. Health economics evaluation index: Average hospital isolation day and cost of hospitalization when patients received treatment, the hospital isolation day is determined by the radiation dose of the patient's body, and the national discharge standard must be met when discharged (400MBq or 25µsv/h).

Data management The original medical records and Case report form（CRF） should be truthfully and carefully recorded as required, and the contents should not be changed easily once filled in. In case of any error, the original record shall not be altered, but shall be supplemented by an additional statement, signed and dated by the physician in charge. All the observed results and abnormal findings in clinical trials should be verified and recorded in time to ensure the reliability of the data. All kinds of instruments, equipment, practice, standard products and so on used in various inspection items in clinical trials should have strict quality standards and ensure that they are working in normal condition.

All data will be programmed with computer software for double input. During this period, the question form will be forwarded to the researcher for data review through the clinical inspector, who should answer and return as soon as possible. The data will be locked by the lead researcher, the applicant, the statistician and the drug supervisor after the blind state audit and think that the established database is correct. No further changes are allowed in the locked data file. The database will be submitted for statistical analysis.

Statistical analysis

1. Statistical software: Statistical Analysis System（SAS）9.4 statistical software is used for statistical analysis.
2. Basic principle: All statistical inferences are performed by two-sided test. The statistically significant test level is set to 0.05, and the confidence interval of the parameters is estimated to be 95% confidence interval. Use the parametric method as much as possible. When the data does not meet the conditions of the parameter method, it can be analyzed by conversion method. If it is still not satisfied, consider using a non-parametric method.
3. Missing data: The integrity of the data is monitored in real time. If the patient is found not to be followed up in time, he will be notified by phone and the data will be filled in time. Withdrawal subjects do not fill in the data.
4. Abnormal data: analysis of causes, exclusion of objective and subjective reasons.
5. Descriptive statistics: The mean number, standard deviation and confidence interval are given in the measurement data. The minimum value, maximum value, P25, median, and P75 are given if necessary; the mean and standard deviation of the difference are given for the paired measurement data; and the median and average rank are given when the non-parametric method is used. The frequency distribution and the corresponding percentage are given by counting data. The frequency distribution and the corresponding percentage, as well as the median number and the average rank, are given. The positive rate, positive number and denominator number are given by qualitative data.
6. analysis of baseline data: descriptive analysis of baseline data (including demographic indicators, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological confirmation of intermediate-risk papillary thyroid carcinoma(PTC) according to 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer.
* Differentiated Thyroid Carcinoma(DTC) patients who underwent total or near-total thyroidectomy which was consistent with the recommendations of American Thyroid Association guidelines as well as Chinese Thyroid Association guidelines on the management of Differentiated Thyroid Carcinoma(DTC).
* Serum stimulated thyroglobulin was 1-20ng/ml.
* At least 16 years old.
* Patients who volunteered to participate in the study and signed informed consent.

Exclusion Criteria:

* Ultrasonography, Computerized Tomography(CT), Magnetic Resonance Imaging(MRI) or Positron Emission Tomography/computed tomography (PET/CT) indicates the presence of lesions.
* Iodine-131 whole body scan indicates the presence of lesions outside the thyroid bed.
* Patients with positive thyroglobulin antibody (≥115 Ku/L).
* Patients who had other coexisting serious diseases or other factors that may affect the outcome of ablation.
* Pregnant or breastfeeding women, or with birth planning within six months.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 3-year
  The 3-years disease-free survival was compared between low-dose group (30 mCi) and high-dose group (100 mCi)

CONTACTS AND LOCATIONS:
Overall Officials: Huijuan Feng, Master, Study Chair — Southern Medical University, China
Locations (1):
- Huijuan Feng, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 12 months of study completion
Access Criteria: Data access requests will be reviewed by an external independent Review Panel

REFERENCES:
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- [Background] Schlumberger M, Catargi B, Borget I, Deandreis D, Zerdoud S, Bridji B, Bardet S, Leenhardt L, Bastie D, Schvartz C, Vera P, Morel O, Benisvy D, Bournaud C, Bonichon F, Dejax C, Toubert ME, Leboulleux S, Ricard M, Benhamou E; Tumeurs de la Thyroide Refractaires Network for the Essai Stimulation Ablation Equivalence Trial. Strategies of radioiodine ablation in patients with low-risk thyroid cancer. N Engl J Med. 2012 May 3;366(18):1663-73. doi: 10.1056/NEJMoa1108586. PMID 22551127
- [Background] Mallick U, Harmer C, Yap B, Wadsley J, Clarke S, Moss L, Nicol A, Clark PM, Farnell K, McCready R, Smellie J, Franklyn JA, John R, Nutting CM, Newbold K, Lemon C, Gerrard G, Abdel-Hamid A, Hardman J, Macias E, Roques T, Whitaker S, Vijayan R, Alvarez P, Beare S, Forsyth S, Kadalayil L, Hackshaw A. Ablation with low-dose radioiodine and thyrotropin alfa in thyroid cancer. N Engl J Med. 2012 May 3;366(18):1674-85. doi: 10.1056/NEJMoa1109589. PMID 22551128
- [Background] Dehbi HM, Mallick U, Wadsley J, Newbold K, Harmer C, Hackshaw A. Recurrence after low-dose radioiodine ablation and recombinant human thyroid-stimulating hormone for differentiated thyroid cancer (HiLo): long-term results of an open-label, non-inferiority randomised controlled trial. Lancet Diabetes Endocrinol. 2019 Jan;7(1):44-51. doi: 10.1016/S2213-8587(18)30306-1. Epub 2018 Nov 27. PMID 30501974